CLINICAL TRIAL: NCT00005178
Title: Study of Children's Activity and Nutrition (SCAN)
Status: Completed | Type: Observational
Sponsor: Augusta University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1056; R01HL035073 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2000-12

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Coronary Disease; Hypertension; Obesity; Hypercholesterolemia; Coronary Heart Disease Risk Reduction
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Coronary Disease; Hypertension; Obesity; Hypercholesterolemia

SUMMARY:
In the first study, to identify children at high and low risk for cardiovascular disease and study their nutritional and physical activity behaviors as they relate to cardiovascular disease. In the second study, to make yearly assessments over a four year period of diet and physical activity among children and their parents. The initial effort redefined and retested methods to collect data on dietary intake and activity levels of young children.

DETAILED DESCRIPTION:
BACKGROUND:

In the past several decades, relationships between various lifestyle behaviors and the development of cardiovascular risk factors have been identified. Nutritional status/eating behaviors and physical activity patterns both directly and indirectly are related to the development of coronary heart disease. For example, obesity, which may be a result of both eating and physical activity behaviors, greatly increases the risk of hypertension, hyperlipidemia, and diabetes mellitus, placing the individuals at greater risk for coronary heart disease. Dietary factors such as composition in fatty acids and cholesterol, composition in vegetable protein and complex carbohydrates, caloric excess and a high intake of salt also are related to the development of risk of coronary heart disease.

Physical activity in adults has also been correlated with coronary heart disease. Epidemiological research has demonstrated that increased physical activity is associated with reduced risk of myocardial infarctions. Regular physical exercise has been shown to have beneficial effects on relative weight and obesity and may act indirectly to beneficially affect hypertension, hypertriglyceridemia and glucose intolerance and raise HDL cholesterol levels. However, in 1985 when SCAN was initiated, little information was available concerning the development of nutritional status/eating behaviors and routine physical activity patterns in children.

Various psychosocial factors have been associated with increased risk of coronary heart disease. Among these factors are behavioral characteristics such as type A behaviors and coping styles to stressors. However, relatively little was known in 1985 concerning the development of such characteristics in children and when these characteristics became associated with risk of cardiovascular disease.

SCAN initiated on the recommendations of the Preventive Cardiology Branch Task Force Group in the Five Year Forward Plan 1982-1987, the Conference on School Health Education Research in the Heart, Lung, and Blood Areas, and the Clinical Applications and Prevention Advisory Committee of the National Heart, Lung, and Blood Institute. A Request for Applications was released in October 1984. In 1985, six grants were awarded as part of the Study of Children's Activity and Nutrition (SCAN).

DESIGN NARRATIVE:

There were six projects supported by the SCAN program. They did not follow a common protocol but were basically similar.

Medical College of Georgia: Five hundred and one Black and white children were followed over a four year period for food intake behavior, physical activity and fitness, anthropometric measurements, blood lipids and lipoproteins, heart rate and blood pressure, and psychologic characteristics associated with coronary heart disease.

West Virginia University: Two hundred and eight predominantly white children of adults followed since adolescence in the Bourbon County Study were members of this cohort. Children participated in cardiovascular fitness tests, and underwent blood pressure measurements, and serum lipid determinations. The effects of television-viewing, child-rearing patterns, exercise, and nutrition-related knowledge and attitudes were assessed over a four year period.

Columbia University: Seven hundred and ninety-four primarily Hispanic children and their parents were followed for four years to determine the extent to which diet and physical activity predict coronary heart disease risk. Cross sectional and longitudinal analyses were performed.

Georgetown University: Five hundred and seventy Black children were followed for the influence of the risk status of an older sibling and day care versus home care on nutrient intake and physical activity. Eating events were videotaped, activity levels were recorded, and measurements were obtained on height, weight, cholesterol, blood pressure, and skinfold thickness. Dietary recalls and nutrition knowledge surveys were obtained.

University of Massachusetts: In the Framingham Children's Study, one hundred children who were direct descendents of Framingham Heart Study participants were followed for four years. Measurements included height, weight, skinfold thickness, lipid profiles, heart rate and activity monitoring, and assessment of dietary intake four times per year.

Memphis State University: Six hundred and sixty-three children and their parents were assessed for food intake, physical activity, and parent-child interactions related to food intake and exercise. Anthropometric and cardiovascular data were also collected every four months for four years.

Two of the studies were renewed in FY 1992 and again in FY 1996. See the Framingham Children's Study and the Children's Activity and Nutrition III.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1985-09; Study Completion 1991-08

CONTACTS AND LOCATIONS:
Overall Officials: R. Ellison; Ronald Iannotti; Robert Klesges; Jane Kotchen; William Strong

REFERENCES:
- [Background] Hulse E, Strong WB. Preparticipation evaluation for athletics. Pediatr Rev. 1987 Dec;9(6):173-82. doi: 10.1542/pir.9-6-173. No abstract available. PMID 3332373
- [Background] Strong WB, Wilmore JH: Unfit Kids: An Office-Based Approach to Physical Fitness. Contemp Pediatr, 4:33-48, 1988
- [Background] Strong WB. So what's good about sports? Am J Dis Child. 1988 Feb;142(2):143. doi: 10.1001/archpedi.1988.02150020041023. No abstract available. PMID 3341313
- [Background] Strong WB, Dennison BA. Pediatric preventive cardiology: atherosclerosis and coronary heart disease. Pediatr Rev. 1988 Apr;9(10):303-14. doi: 10.1542/pir.9-10-303. No abstract available. PMID 3054834
- [Background] Strong WB (Ed): In: The Pediatrician of the 90's. Biomedical Information Corporation, 1988
- [Background] Arensman FW, Treiber FA, Gruber MP, Strong WB. Exercise-induced differences in cardiac output, blood pressure, and systemic vascular resistance in a healthy biracial population of 10-year-old boys. Am J Dis Child. 1989 Feb;143(2):212-6. doi: 10.1001/archpedi.1989.02150140106030. PMID 2916494
- [Background] Treiber FA, Musante L, Strong WB, Levy M. Racial differences in young children's blood pressure. Responses to dynamic exercise. Am J Dis Child. 1989 Jun;143(6):720-3. doi: 10.1001/archpedi.1989.02150180102029. PMID 2729217
- [Background] Treiber FA, Musante L, Hartdagan S, Davis H, Levy M, Strong WB. Validation of a heart rate monitor with children in laboratory and field settings. Med Sci Sports Exerc. 1989 Jun;21(3):338-42. PMID 2733584
- [Background] Treiber FA, Mabe PA 3rd, Riley W, Carr T, Levy M, Thompson W, Strong WB. Assessment of children's Type A behavior: relationship with negative behavioral characteristics and children and teacher demographic characteristics. J Pers Assess. 1989 Winter;53(4):770-82. doi: 10.1207/s15327752jpa5304_13. PMID 2607405
- [Background] Musante L, Treiber FA, Strong WB, Levy M. Family history of hypertension and cardiovascular reactivity to forehead cold stimulation in black male children. J Psychosom Res. 1990;34(1):111-6. doi: 10.1016/0022-3999(90)90014-u. PMID 2313609
- [Background] Strong WB. Physical activity and children. Circulation. 1990 May;81(5):1697-701. doi: 10.1161/01.cir.81.5.1697. No abstract available. PMID 2184948
- [Background] Musante L, Treiber FA, Strong WB, Levy M. Individual and cross-spouse correlations of perceptions of family functioning, blood pressure and dimensions of anger. J Psychosom Res. 1990;34(4):393-9. doi: 10.1016/0022-3999(90)90062-9. PMID 2376840
- [Background] Segal KR, Gutin B, Presta E, Wang J, Van Itallie TB. Estimation of human body composition by electrical impedance methods: a comparative study. J Appl Physiol (1985). 1985 May;58(5):1565-71. doi: 10.1152/jappl.1985.58.5.1565. PMID 3997721
- [Background] Gutin B, Alejandro D, Duni T, Segal K, Phillips GB. Levels of serum sex hormones and risk factors for coronary heart disease in exercise-trained men. Am J Med. 1985 Jul;79(1):79-84. doi: 10.1016/0002-9343(85)90549-2. PMID 3893124
- [Background] Gutin B: Basic Principles of Training and Fitness. Contemporary OB/GYN. Special Issue on The Active Women, May 1985
- [Background] Segal KR, Gutin B, Nyman AM, Pi-Sunyer FX. Thermic effect of food at rest, during exercise, and after exercise in lean and obese men of similar body weight. J Clin Invest. 1985 Sep;76(3):1107-12. doi: 10.1172/JCI112065. PMID 4044828
- [Background] Michela JL, Contento IR. Cognitive, motivational, social, and environmental influences on children's food choices. Health Psychol. 1986;5(3):209-30. doi: 10.1037//0278-6133.5.3.209. PMID 3743530
- [Background] Gutin B, Gutin C: Obesity Prevention and Exercise in Countries Undergoing Technological Development. Physician & Sportsmedicine, 14(10):197-201, 1986
- [Background] Segal KR, Gutin B, Albu J, Pi-Sunyer FX. Thermic effects of food and exercise in lean and obese men of similar lean body mass. Am J Physiol. 1987 Jan;252(1 Pt 1):E110-7. doi: 10.1152/ajpendo.1987.252.1.E110. PMID 3812669
- [Background] Gutin B, Mayers M, Levy J, Herman M: Physiologic & Echocardiographic Studies of Age-Group Runners. In: Brown E (Ed) Competitive Sports for Children & Youths. Champaign: Human Kinetics, 1987
- [Background] DeLozier M, Gutin B, Wang J, Zybert P, Basch C, Rips J, Shea S, Contento I, Irigoyen M, Pierson R: Bio-Impendance Derived Estimates of Body Composition in 4-8 Years Olds. Medicine and Science in Sports and Exercise, 20:S31, 1988
- [Background] Shea S, Basch CE, Zybert P, Rips J, Contento I, Gutin B, Irigoyen M. Screening using National Cholesterol Education Program guidelines in a population of urban Hispanic mothers. Prev Med. 1989 Nov;18(6):824-32. doi: 10.1016/0091-7435(89)90018-2. PMID 2626415
- [Background] Shea S, Basch CE, Irigoyen M, Zybert P, Rips JL, Contento I, Gutin B. Failure of family history to predict high blood cholesterol among hispanic preschool children. Prev Med. 1990 Jul;19(4):443-55. doi: 10.1016/0091-7435(90)90042-i. PMID 2204914
- [Background] Basch CE. Focus group interview: an underutilized research technique for improving theory and practice in health education. Health Educ Q. 1987 Winter;14(4):411-48. doi: 10.1177/109019818701400404. PMID 3319971
- [Background] DeLozier M, Rips J, Gutin B, and Basch C: Strategies and Techniques for Conducting Treadmill Tests in Preschool-Age Children, J Phys Educ, Recreat and Dance, forthcoming, 1988
- [Background] Ellison RC: Dangers of Screening for Hyperlipidemia in Children (letter to the editor). N Engl J Med, 314:1579-1580, 1986
- [Background] Witschi JC, Capper AL, Hosmer DW Jr, Ellison RC. Sources of sodium, potassium, and energy in the diets of adolescents. J Am Diet Assoc. 1987 Dec;87(12):1651-5. PMID 3680823
- [Background] Ellison RC. Give diet a chance in lowering cholesterol levels. Arch Intern Med. 1988 May;148(5):1017-9. No abstract available. PMID 3365070
- [Background] Klesges LM, Klesges RC. The assessment of children's physical activity: a comparison of methods. Med Sci Sports Exerc. 1987 Oct;19(5):511-7. PMID 3683156
- [Background] Klesges RC, Klesges LM, Brown G, Frank GC. Validation of the 24-hour dietary recall in preschool children. J Am Diet Assoc. 1987 Oct;87(10):1383-5. PMID 3655169
- [Background] Klem ML, Klesges RC. Competition in a minimal-contact weight-loss program. J Consult Clin Psychol. 1988 Feb;56(1):142-4. doi: 10.1037//0022-006x.56.1.142. No abstract available. PMID 3346440
- [Background] Weber JM, Klesges RC, Klesges LM. Dietary restraint and obesity: their effects on dietary intake. J Behav Med. 1988 Apr;11(2):185-99. doi: 10.1007/BF00848265. PMID 3172191
- [Background] Myers RJ, Klesges RC, Eck LH, Hanson CL, Klem ML. Accuracy of self-reports of food intake in obese and normal-weight individuals: effects of obesity on self-reports of dietary intake in adult females. Am J Clin Nutr. 1988 Nov;48(5):1248-51. doi: 10.1093/ajcn/48.5.1248. PMID 3189212
- [Background] Klesges RC, Hanson CL, Eck LH, Durff AC. Accuracy of self-reports of food intake in obese and normal-weight individuals: effects of parental obesity on reports of children's dietary intake. Am J Clin Nutr. 1988 Nov;48(5):1252-6. doi: 10.1093/ajcn/48.5.1252. PMID 3189213
- [Background] Eck LH, Klesges RC, Hanson CL. Recall of a child's intake from one meal: are parents accurate? J Am Diet Assoc. 1989 Jun;89(6):784-9. PMID 2723300
- [Background] Cohen R, Klesges RC, Summerville M, Meyers AW. A developmental analysis of the influence of body weight on the sociometry of children. Addict Behav. 1989;14(4):473-6. doi: 10.1016/0306-4603(89)90036-1. PMID 2675542
- [Background] Klesges RC, Meyers AW, Klesges LM, La Vasque ME. Smoking, body weight, and their effects on smoking behavior: a comprehensive review of the literature. Psychol Bull. 1989 Sep;106(2):204-30. doi: 10.1037/0033-2909.106.2.204. PMID 2678202
- [Background] Williams E, Klesges RC, Hanson CL, Eck LH. A prospective study of the reliability and convergent validity of three physical activity measures in a field research trial. J Clin Epidemiol. 1989;42(12):1161-70. doi: 10.1016/0895-4356(89)90114-5. PMID 2585007
- [Background] Mizes JS, Klesges RC. Validity, reliability, and factor structure of the Anorectic Cognitions Questionnaire. Addict Behav. 1989;14(5):589-94. doi: 10.1016/0306-4603(89)90081-6. PMID 2589139
- [Background] Klesges RC, Klem ML, Bene CR. Effects of dietary restraint, obesity, and gender on holiday eating behavior and weight gain. J Abnorm Psychol. 1989 Nov;98(4):499-503. doi: 10.1037//0021-843x.98.4.499. PMID 2592685
- [Background] Klesges RC, Eck LH, Isbell TR, Fulliton W, Hanson CL. Smoking status: effects on the dietary intake, physical activity, and body fat of adult men. Am J Clin Nutr. 1990 May;51(5):784-9. doi: 10.1093/ajcn/51.5.784. PMID 2333836
- [Background] Klem ML, Klesges RC, Bene CR, Mellon MW. A psychometric study of restraint: the impact of race, gender, weight and marital status. Addict Behav. 1990;15(2):147-52. doi: 10.1016/0306-4603(90)90018-s. PMID 2343788
- [Background] Klesges RC, Haddock CK, Eck LH. A multimethod approach to the measurement of childhood physical activity and its relationship to blood pressure and body weight. J Pediatr. 1990 Jun;116(6):888-93. doi: 10.1016/s0022-3476(05)80645-6. PMID 2348291
- [Background] Klesges RC, Eck LH, Hanson CL, Haddock CK, Klesges LM. Effects of obesity, social interactions, and physical environment on physical activity in preschoolers. Health Psychol. 1990;9(4):435-49. doi: 10.1037//0278-6133.9.4.435. PMID 2373068
- [Background] Klesges RC, Klem ML, Hanson CL, Eck LH, Ernst J, O'Laughlin D, Garrott A, Rife R. The effects of applicant's health status and qualifications on simulated hiring decisions. Int J Obes. 1990 Jun;14(6):527-35. PMID 2401589
- [Background] Treiber FA, Musante L, Braden D, Arensman F, Strong WB, Levy M, Leverett S. Racial differences in hemodynamic responses to the cold face stimulus in children and adults. Psychosom Med. 1990 May-Jun;52(3):286-96. doi: 10.1097/00006842-199005000-00003. PMID 2367620
- [Background] DuRant RH, Baranowski T, Rhodes T, Gutin B, Thompson WO, Carroll R, Puhl J, Greaves KA. Association among serum lipid and lipoprotein concentrations and physical activity, physical fitness, and body composition in young children. J Pediatr. 1993 Aug;123(2):185-92. doi: 10.1016/s0022-3476(05)81687-7. PMID 8345412